CLINICAL TRIAL: NCT03431922
Title: Endovascular Denervation in Patients With Cancer Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Dean, Zhongda Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ED treatment
Record Dates: First submitted 2018-01-19; First posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Cancer Pain
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- endovascular denervation (Experimental): endovascular denervation
  Interventions: Device: endovascular denervation

INTERVENTIONS:
Device: endovascular denervation — multi-electrode catheter-based endovascular denervation

SUMMARY:
Endovascular arterial denervation (ED) is a minimally invasive technique which could reduce the occurrence of injury of visceral tissue or organs. As the principle of renal denervation (RDN), Radiofrequency energy delivered by a multi-electrode catheter to the celiac plexus over the anterolateral surface of the superior mesenteric artery (SMA) and the celiac axis. Damaged or partially damaged celiac plexus can achieve the effect of pain relief.

DETAILED DESCRIPTION:
The multi-electrode catheter was consisted of six independent electrodes helically on a net structure, which could be set as the same energy and temperature for simultaneous multi-point ablation. A real-time monitoring capability also provided by the display.

ELIGIBILITY:
Inclusion Criteria:

* 25 to 75 years
* severe cancer pain with the visual analogue scores of no less than 7

Exclusion Criteria:

* pregnant or intent to become pregnant within 1 year
* postural hypotension
* uncorrected coagulation dysfunction
* aortic aneurysm or dissection
* type 1 diabetes mellitus (T1DM)
* acute or severe systemic infection
* history of cerebral apoplexy or transient ischemic attack (TIA) in the past two weeks
* history of acute coronary syndrome in the past two weeks
* participants who are not suitable to be enrolled into the study assessed by the researchers

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-09-21 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Pain relief | from baseline to 1 months after procedure
  Changes of the visual analogue scores (VAS) scores

SECONDARY OUTCOMES:
Pain relief | from baseline to 3 months after procedure
  Changes of the visual analogue scores (VAS) scores
Improvement of Quality of Life | from baseline to 3 months after procedure
  Changes of the 100-item World Health Organization Quality of Life (QOL)
Incidence of Treatment Adverse Events | from baseline to 1 months after procedure
  Assess artery damage, such as abdominal aortic dissection and abdominal aneurysm, by digital subtraction angiography or computed tomography

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, MD, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Oliveira R, dos Reis MP, Prado WA. The effects of early or late neurolytic sympathetic plexus block on the management of abdominal or pelvic cancer pain. Pain. 2004 Jul;110(1-2):400-8. doi: 10.1016/j.pain.2004.04.023. PMID 15275792
- [Background] Wong GY, Schroeder DR, Carns PE, Wilson JL, Martin DP, Kinney MO, Mantilla CB, Warner DO. Effect of neurolytic celiac plexus block on pain relief, quality of life, and survival in patients with unresectable pancreatic cancer: a randomized controlled trial. JAMA. 2004 Mar 3;291(9):1092-9. doi: 10.1001/jama.291.9.1092. PMID 14996778
- [Background] Cleeland CS, Gonin R, Hatfield AK, Edmonson JH, Blum RH, Stewart JA, Pandya KJ. Pain and its treatment in outpatients with metastatic cancer. N Engl J Med. 1994 Mar 3;330(9):592-6. doi: 10.1056/NEJM199403033300902. PMID 7508092